CLINICAL TRIAL: NCT05093218
Title: Effect of Branch Chain Amino Acid Therapy on Sarcopenia in Children With Chronic Liver Disease-A Double Blinded RCT
Brief Title: Effect of Branch Chain Amino Acid Therapy on Sarcopenia in Children With Chronic Liver Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-CLD-03
Record Dates: First submitted 2021-09-27; First posted 2021-10-26 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-09

CONDITIONS: Sarcopenia; Cirrhosis, Liver
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- branch chain amino acid (Experimental): • Branch chain amino acid at a dose of approxiametely 0.35g/kg will be supplemented in two divided doses group for a period of 12 weeks.For the sake of administration, it will be prescribed as per the following weight band categories: <5kg 2 gm 5-10kg 4 gm 10-20kg 8 gm 20-40kg 12 gm 40-60kg 24 gm
  Interventions: Dietary Supplement: branch chain amino acid
- placebo (Placebo Comparator): Placebo will have the similar colour, taste and consistency. Both groups will be given the same dose.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: branch chain amino acid — • Branch chain amino acid at a dose of approxiametely 0.35g/kg will be supplemented in two divided doses group for a period of 12 weeks.For the sake of administration, it will be prescribed as per the following weight band categories: <5kg 2 gm 5-10kg 4 gm 10-20kg 8 gm 20-40kg 12 gm 40-60kg 24 gm
  Arms: branch chain amino acid
Other: placebo — Placebo will have the similar colour, taste and consistency. Both groups will be given the same dose.
  Arms: placebo

SUMMARY:
Sarcopenia is now a well-known complication of cirrhosis and various studies, including pediatric studies, have recognized it as a poor prognostic factor. At the molecular level, branch chain amino acids upregulate muscle protein synthesis by acting through the mTOR pathway. Although effect of Branch Chain Amino acids has been studied extensively with respect to hepatic encephalopathy in cirrhotic adults, there is paucity of literature on the effect of BCAA on sarcopenia and frailty. Also, there is very limited data on the effect of BCAA therapy in children with chronic liver disease. Through this study, we aim to assess the effect of BCAA therapy on Mid Arm Muscle Area in cirrhotic children after 12 weeks. Our secondary objective will be to study the prevalence of sarcopenia in children with CLD using cut-off as Mid Arm Muscle area less than 2SD (using published centiles) and muscle thickness (quadriceps and biceps) on ultrasound, and to study serum follistatin levels in those with or without sarcopenia. Other secondary objectives will include determination of mTOR gene expression at baseline and 7 days of BCAA therapy and change in creatinine height index after 12 weeks of BCAA therapy, occurrence of clinically significant events in the BCAA group vs placebo group and to study the increase in MAMA and USG muscle thickness after 6 months of BCAA therapy.

DETAILED DESCRIPTION:
Study Design: Single centre randomized double blinded placebo Control Trial.

Primary objective:

To assess increase in Mid-arm muscle area (MAMA) after 12 weeks of BCAA therapy in children with CLD and sarcopenia (MAMA <2 SD).

Secondary objectives:

To study the

* Prevalence of Sarcopenia defined by MAMA <2SD for age in children with cirrhosis.
* Prevalence of sarcopenia based on USG muscle size (biceps and quadriceps) in children with cirrhosis.
* Follistatin levels in children with CLD with and without sarcopenia.
* Change in mTOR gene expression levelsafter 7 days of BCAA therapy.
* Change in creatinine-height index after 12 weeks of BCAA therapy.
* Change in MAMA (muscle size) after 6 months of BCAA therapy.
* Change in muscle size (biceps and quadriceps) using ultrasound at 3 and 6 months.
* Occurrence of significant events including HE, UGI bleed, SBP, AKI, new onset or increase in ascites, hospital stay and mortality in the BCAA group versus placebo at 3 and 6 months.
* Albumin requirement over 3 and 6 months.

Study population:

Children with cirrhosis with Sarcopenia (6 mo - 12 years) fulfilling the conditions as per inclusion and exclusion criteria.

Baseline parameters that will be recorded:

Clinical parameters: Jaundice, Organomegaly, HE(overt and minimal), ascites, SBP, cholangitis , upper GI bleed, AKI Laboratory parameters: Complete blood count, LFT, KFT, PT-INR, ammonia, mTOR gene expression, serum follistatinlevel, 24hr urine creatinine Imaging parameters: Splenic size on USG, Splenic Z-score, PV diameter, USG muscle - biceps and quadriceps

Anthropometric parameters:

Weight for age Height for age Triceps skin fold thickness Subscapular skin fold thickness Mid arm circumference MAMC calculated as MUAC-(TSF*3.14) MAMA calculated as (MUAC-(〖3.14*TSF)〗^2)/(4*3.14)

Calculation of Sarcopenia cut-off:

Cut-off for sarcopenia will be defined as Mid Arm Muscle area less than 2 SD based on MAMA centiles of normal healthy American children as studied by Addo OY et al.

Methodology for USG for muscle thickness:

Ultrasound scans, both baseline and at follow-up, will be done in the same setting with the participant in supine lying position with the knee fully extended, hip in a neutral position and ankles relaxed in a slight plantar flexion for the lower limb and arm fully extended for the upper limb.

Muscle Site of measurement Definition of muscle thickness Biceps brachii Two third of distance from acromion to antecubital crease Distance between humerus and ventral fascia of biceps

Quadriceps One half of distance between ASIS and superior aspect of patella Distance between femur and ventral fascia of rectus femoris

The site of measurement will be as follows:

The scanning site will be marked with a skin-marking pen. The transducer will be coated with a generous amount of ultrasound water-based transmission gel and placed perpendicular to the skin applying the lightest contact pressure to ensure that underlying tissues are not compressed. Scanner parameters will remain the same for all measurements, ensuring uniformity to the baseline measurements procedure. Three consecutive readings will be recorded.

The cut-off for normal muscle thickness will be taken from the following formula provided by Scholten RR et al:

Normal biceps brachii muscle thickness (in cm) = 0.77+0.028*weight (SD 0.16) Normal quadriceps muscle thickness (in cm) = 1.63+0.042* weight( SD 0.34) To look for inter-observer variation in assessing muscle size on Ultrasound, this will be done by 2 persons for around 50% of observations in the study.

Alongwith routine investigations including Complete Blood counts, Liver function and Renal function test, PT-INR, serum Ammonia, the following investigations will also be done:

Serum follistatin levels at baseline: This will be done with kit-based ELISA.

mTOR gene expression at baseline and at Day 7: 1 ml blood will be drawn in EDTA vial. The total RNA will be isolated by Trozol RNA isolation protocol. Further these isolated RNAs will be reverse transcribed by CDNA kit. Following this, Real time PCR will be performed in the presence of SYBER Green fluorescent dye. Reverse primers of targeted genes of mTOR-pathway includes p-mTOR (Ser2448), mTOR, p-Akt (Thr308), Akt, Nrf2, UCP-2 (C-terminal) p-AMPK (Thr172 or Ser485/491) and AMPK, p-p65. GAPDH, a housekeeping gene, will be used as a normalization control. The thermal cycling conditions will be 10 min 95°C, followed by 40 cycles of 15 sec at 95°C and 1 min at 60°C. Each measurement will be performed in triplicate and relative gene expression will be determined by the ∆CT method. The same process will be done in the blood samples procured after 7 days of BCAA therapy.

Creatinine height index at baseline and at 12 weeks: This will be calculated as per the following formula(24 hour urine creatine)/(Expected 24 hr urine creatinine for same sex andheight)

Following enrolment and those fulfilling inclusion criteria, patient will then be allocated into BCAA or placebo group as per block randomization method and there will be allocation-concealment with sealed 4 digit and coded envelopes. BCAA or placebo will be supplemented for a period of 12 weeks. Patient will be followed up for a period of 12 weeks. At the end of 12 weeks, mid arm muscle circumference will be repeated. USG muscle thickness, routine blood investigations, creatinine height index will also be repeated. mTOR gene expression will be repeated at 7 days.

Occurrence of clinical events including new onset ascites, AKI, hepatic encephalopathy, upper GI bleed and overall hospital stay as well as mortality over 12 weeks and 6 months will be noted in both groups during this period and treated as per standard of care. These events will be defined as follows- Acute Kidney Injury

As per KDIGO guidelines:

Increase in serum creatinine by more than 0.3mg/dl within 48 hours, OR Urine output less than 0.5ml/kg/hour for more than 6 hours, OR Increase in serum creatinine by more than 1.5 times the baseline presumed/known to have occurred within prior 7 days.

Hepatic encephalopathy: as per Modified West-Haven's criteria.

Grades of ascites Grade 1- ascites only detected by ultrasound Grade 2 -moderate ascites evident by distension of abdomen with shifting dullness Grade 3- gross/tense ascites with marked abdominal distension

Study period: 2 years

Sample size with justification:

Observational part: Assuming prevalence of sarcopenia in children with chronic liver disease is 40%, with alpha of 5%, permissible error of 10%, we need to enroll 96 cases to estimate the prevalence of sarcopenia in children with CLD.

Interventional (RCT part): Assuming that baseline MAMC values in BCAA and control group are same, after follow up of 3 months, the MAMC value in BCAA by a value of 4.6 cm (18% change, 30.5 vs 25.9 cm) (Ruiz-Margain A et al, Rev de Gastroenterol de Mexico 2018) with alpha -5% and power of 90%, we need to enroll total 40 cases. Assuming attrition rate of 10%, it was decided to enroll 44 cases randomly allocated into 2 groups by block randomisation method with block size of 4.

Intervention:

Branch chain amino acid at a dose of approxiametely 0.35g/kg will be supplemented in two divided doses group for a period of 12 weeks.For the sake of administration, it will be prescribed as per the following weight band categories:

<5kg 2 gm 5-10kg 4 gm 10-20kg 8 gm 20-40kg 12 gm 40-60kg 24 gm Placebo will have the similar colour, taste and consistency. Both groups will be given the same dose.

Both groups will be advised a calorie intake of 150cal/kg/day and protein intake of 2-2.5gm/kg/day, and this will be ensured in regular follow-up as a standard care of practice developed by the department of Pediatric Hepatology.

Monitoring and assessment:

Patients will be followed up for a period of at least 6 months. Occurrence of clinical events including new onset ascites, AKI, hepatic encephalopathy, upper GI bleed, significant infections will be noted in both groups during this period and treated as per standard of care.

At the end of 12 weeks, mid arm muscle circumference and other anthropometric parameters, muscle thickness on ultrasonography, and creatinine height index will also be repeated. mTOR gene expression will be repeated at the end of 7 days. Mid arm muscle circumference and other anthropometric parameters, and muscle thickness on ultrasonography will again be repeated at 6 months.

Statistical Analysis All the categorical variables will be expressed as frequencies, whereas continuous ones will be expressed as mean or median ± SD. Chi-square test and student's t-test (Fisher's exact test) will be applied for assessment of causality. Kaplan-Meyer statistics will be done for survival and liver related morbidity. Significance will be mentioned in the form of p-value <0.05 and as Odd's ratio and 95% confidence interval.

Adverse effects:

There are no expected adverse effects of Branch chain amino acids as seen in previous studies.

Stopping rule of study:

Interruption of supplementation for 15 consecutive days due to non-compliance or clinical events.

Progression to exclusion criteria i.e. development of malignancy, AKI, potential liver transplant within 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 mo - 12 y with cirrhosis and sarcopenia defined as MAMA <2 SD for age

Exclusion Criteria:

1. Non-cirrhotic Portal hypertension
2. Suspected/proven malignancy
3. Already on BCAA therapy in last 1 month
4. Tyrosinemia
5. Chronic kidney disease or non-resolving AKI
6. Potential liver transplant within 1 month.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2021-10-31 (Actual); Primary Completion 2023-03-05 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Change in Mid-arm muscle area (MAMA) after 12 weeks of BCAA therapy in children with CLD and sarcopenia (MAMA <2 SD). | 12 weeks
  Mid-arm Muscle area (MAMA) is a measure of sarcopenia (muscle mass) and this we are assessing to know whether Branched chain amino-acid supplementation will influence muscle mass at 12 weeks. MAMA will be calculated from triceps skin fold thickness and Mid arm circumference using the formula, MAMA = [(MAC - 3.14*TSF)^2]/4*3.14

SECONDARY OUTCOMES:
Change in mTOR gene expression levels after 7 days of BCAA therapy | 7 days
Change in follistatin levels in children with CLD after 12 weeks of BCAA therapy. | 12 weeks
Change in creatinine-height index after 12 weeks of BCAA therapy. | 12 weeks
Change in MAMA (muscle size) after 6 months of BCAA therapy. | 6 months
Change in muscle size (biceps and quadriceps) using ultrasound at 3 and 6 months. | 3 months
Change in muscle size (biceps and quadriceps) using ultrasound at 3 and 6 months. | 6 months
Change in Albumin requirement over 3 and 6 months in the BCAA group | 3 months
Change in Albumin requirement over 3 and 6 months in the BCAA group | 6 months
Change in the occurrence of significant events including HE, UGI bleed, SBP, AKI, new onset or increase in ascites, hospital stay and mortality in the BCAA group versus placebo at 3 and 6 months. | 3 months
Change in the occurrence of significant events including HE, UGI bleed, SBP, AKI, new onset or increase in ascites, hospital stay and mortality in the BCAA group versus placebo at 3 and 6 months. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institiute of liver and biliary sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided